CLINICAL TRIAL: NCT04043130
Title: The Evaluation of Pulse: A Mobile Health App and Teen Pregnancy Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Child Trends (Other)
Collaborators: Healthy Teen Network (Other); Ewald and Wasserman (Unknown); MetaMedia Training International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TP2AH000038
Record Dates: First submitted 2019-03-01; First posted 2019-08-02 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Unprotected Sex; Contraceptive Usage
Keywords: Reproductive and Sexual Health Care Utilization
MeSH Terms: conditions — Unsafe Sex; Contraception Behavior | interventions — Pulse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulse Treatment App (Experimental): The treatment app is a web-based mobile health app designed for Black & Latinx women ages 18-20. Through culturally and age-appropriate content, Pulse provides information on birth control, healthy relationships, sexual health, pregnancy, & utilization of clinical services to encourage users to choose effective birth control, seek reproductive health services, and prevent unplanned pregnancies. Users access Pulse autonomously and on their own terms. The app does not require users to follow a specific sequence of content viewed. Participants randomized to the intervention condition are given access to Pulse and receive Multimedia Messaging Service (MMS) messages related to sexual health several times a week for 6 weeks. Participants receive a baseline survey, 6-week follow-up survey, and 6-month follow-up survey via an electronic survey platform (6-month survey only administered to participants recruited between November 2018-March 2019).
  Interventions: Behavioral: Pulse
- Pulse Control App (Active Comparator): The control app, also called Pulse, is a web-based mobile health app designed by the study team for young women ages 18-20. Although Pulse control and Pulse treatment apps look and feel similar aesthetically, they contain different content. Pulse control app provides information on general health topics, such as the importance of sleep, healthy eating, and friendships. Users access Pulse autonomously, on their own terms, and in their own time and place. The app does not require the user to follow a specific sequence of content viewed; however, all users receive a monetary incentive after completing a baseline survey and registering with the app. Control participants also receive MMS messages related to general health for six weeks. Participants receive a baseline survey and a six-week follow-up which are conducted online via an electronic survey platform.
  Interventions: Behavioral: Pulse

INTERVENTIONS:
Behavioral: Pulse — The intervention provides participants access to Pulse, a web-based mobile health app designed for Black and Latinx women ages 18-20. Participants can access the app autonomously and on their own schedule. The app for the experimental arm, the Pulse treatment app, provides information on birth control, healthy relationships, sexual health and physiology, pregnancy, and utilization of clinical services. The app for the comparator arm, the Pulse control app, provides information on general health topics, such as the importance of sleep, healthy eating, and friendships. Participants receive MMS messages that reinforce app content and remind them to visit the app.
  Other Names: GirlPower

SUMMARY:
This study used a randomized controlled design to evaluate the efficacy of a new mobile app, Pulse, in reducing the incidence of unprotected sex among young women. Pulse is a web-based mobile health application that can be accessed through mobile smartphones and computers. Pulse was designed to increase highly effective birth control use and reproductive and sexual health care utilization, and ultimately decrease teen pregnancy. The sample was comprised of 2,317 women aged 18-20 who, at enrollment, were not pregnant or trying to become pregnant, had daily access to a smartphone, were currently living in the United States or a U.S. territory, and spoke English. Most of the sample (86%) identified as Black and/or Latinx. The evaluation team enrolled participants over a two and a half year enrollment period using social media, including Facebook and Instagram.

Users accessed Pulse autonomously, on their own terms, and in their own time and place. The app consists of 6 sections and includes 3 hours of unique content. It does not require the user to follow a specific sequence of content viewed; however, all users received a monetary incentive after registering with the app. Young women randomized to the intervention condition were given access to Pulse indefinitely and received daily text messages related to sexual health for 6 weeks. Control participants were directed to a free general health/fitness web-based mobile application, also called Pulse, and received text messages related to general health for 6 weeks. The control and treatment apps look and feel similar aesthetically but contain different content. Participants in both the intervention and comparison groups received a baseline survey, a 6-week follow-up survey, and a 6-month follow-up survey (the 6-month follow-up survey was only administered to participants recruited between November 2018 and March 2019). Participants also received incentives for completing the baseline and post-intervention surveys. Both surveys were conducted online via an electronic survey platform. This study was conducted as a Rigorous Evaluation of New or Innovative Approaches to Prevent Teen Pregnancy funded by the U.S. Department of Health and Human Services' Office of Adolescent Health.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Female
* Age Limit: 18-20
* Must have daily access to a smartphone that receives text messages and can access the Internet
* Must speak English
* Must live in the United States or a U.S. territory

Exclusion Criteria:

* Currently pregnant or trying to get pregnant

Ages: 18 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 2317 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Unprotected sex, no contraceptive | Baseline (unprotected sex in the past 3 months)
  Ever having sexual intercourse without using any method of contraception (among full sample)
Unprotected sex, no contraceptive | 6-week post-baseline (in the past 6 weeks)
  Ever having sexual intercourse without using any method of contraception (among full sample)
Unprotected sex, no contraceptive | 6-months post-baseline (in the past 3 months)
  Ever having sexual intercourse without using any method of contraception (among full sample)
Unprotected sex, no highly effective contraceptive | Baseline (unprotected sex in the past 3 months)
  Ever having sexual intercourse without using a hormonal or LARC method of contraception (among full sample)
Unprotected sex, no highly effective contraceptive | 6-week post-baseline (in the past 6 weeks)
  Ever having sexual intercourse without using a hormonal or LARC method of contraception (among full sample)
Unprotected sex, no highly effective contraceptive | 6-months post-baseline (in the past 3 months)
  Ever having sexual intercourse without using a hormonal or LARC method of contraception (among full sample)

SECONDARY OUTCOMES:
Reproductive and sexual health care utilization (among full sample) | 6-week post-baseline (in the past 6 weeks)
  Visiting a health care provider for reproductive or sexual health services within the past 6 weeks for the 1st follow-up survey
Reproductive and sexual health care utilization (among full sample) | 6-months post-baseline (in the past 6 months)
  Visiting a health care provider for reproductive or sexual health services within the past 6 months for the 1st follow up survey

CONTACTS AND LOCATIONS:
Locations (1):
- Healthy Teen Network, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No